CLINICAL TRIAL: NCT01125098
Title: Comparison of a Serum Procalcitonin (PRO-CT) Guided Treatment Plan With the Standard Guideline Recommended Antibiotic Treatment Plan for Patients Hospitalized With a Diagnosis of Exacerbation of COPD
Brief Title: Comparison of a Serum PRO-CT Guided Treatment and the Recommended Antibiotic Treatment for COPD
Status: Completed | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Principal Investigator, Leonardo M. Fabbri, Professor Medical Doctor, University of Modena and Reggio Emilia
Other Study IDs: FARM58J2XH
Record Dates: First submitted 2010-04-13; First posted 2010-05-18 (Estimated); Results first posted 2014-12-17 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; PRO-CT; antibiotics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Amoxicillin; Clavulanic Acid; Quinolones

STUDY DESIGN:
Biospecimen Retention: Samples Without DNA — Blood samples and sputum will be collected from COPD patients in order to measure serum PRO-CT levels and inflammatory markers (cells and mediators), respectively.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PRO-CT group: Experimental: COPD patients in the PRO-CT group will continue or discontinue antibiotic therapy depending on PRO-CT values.
  Interventions: Other: PRO-CT values
- Standard group: No intervention: COPD patients in the Standard group will continue antibiotic therapy for 10 days according to guidelines recommended treatment plan in case of COPD exacerbations.

INTERVENTIONS:
Other: PRO-CT values — * continue antibiotics for 10 days if a single PRO-CT value is 0.25 mcg/L or greater, that will be judged suggestive of bacterial infection
  * continue antibiotics from day 3 to day 10 if one or more PRO-CT values are 0.1 to 0.25 mcg/L, indicative of possible bacterial infection, PLUS acute respiratory failure or clinical instability
  * stop antibiotics on day 3, if one or more PRO-CT values are between 0.1 to 0.25 mcg/L, indicative of possible bacterial infection, BUT the patient has not acute respiratory failure or clinical instability
  * stop antibiotics if all the PRO-CT values are < 0.1 mcg/L or if there is a consistent trend to normalization of PRO-CT with the last value < 0.1 mcg/L, that will be judged suggestive of absence of bacterial infection.
  Other Names: Amoxicilline + Clavulanate OR Quinolones
  Groups: PRO-CT group: Experimental

SUMMARY:
Exacerbations of chronic obstructive pulmonary disease (COPD) are the first cause of admission to Pulmonary Department in Italy and worldwide. Guidelines recommend treating most patients hospitalized for exacerbations of COPD with antibiotics, even if the role of bacterial infection is often uncertain and the effect of antibiotics poor. The recommendation to use antibiotics is guided by clinical signs and symptoms that have an insufficient diagnostic accuracy, whereas serum biomarkers as procalcitonin (PRO-CT) may guide the selection of COPD patients who need antibiotic treatment. The main aim of the study is to investigate whether antibiotics can be safely stopped after 3 days or continued for 10 days according to a PRO-CT-guided algorithm in patients hospitalized for exacerbations of COPD for whom guidelines recommend 3-10 days antibiotic treatment based on presence of increased dyspnoea, sputum and purulence. The study is designed to assess the non inferiority of the PRO-CT guided plan as compared to the standard guideline recommended plan. The PRO-CT guided withholding of antibiotics is viewed as an experimental intervention associated with less antibiotic-associated complications, eg antibiotic resistance and drug-related side-effect and lower costs. The proposed study is a prospective, randomised controlled, single-blinded intervention trial comparing the standard with a PRO-CT guided antibiotic treatment plan. Patients will be recruited from the Pulmonary Department of 18 University or City Hospitals in Italy, starting October 2006 and continuing until December 2010. Results expected by end of 2011. The 100 patients randomised to the standard non PRO-CT guided antibiotic treatment plan will continue antibiotics for 10 days, whereas the 100 patients randomised to the PRO-CT guided antibiotic treatment plan will continue for 10 days or stop antibiotics on day 3 depending on PRO-CT levels measured at admission, day 1 and day 2. Serum PRO-CT will be measured in a central laboratory. Patients will be examined at admission, discharge, 10 days, 1, 3 and 6 months. A telephone interview will be obtained at 2, 4 and 5 months. The primary outcome of the study will be the rate of exacerbations. Secondary outcomes will be hospital readmission, admission to ICU, change in FEV1, duration of hospitalization, and death. The sample size was estimated according to the primary outcome of the study.

DETAILED DESCRIPTION:
Patients will be recruited from the Pulmonary Department of 18 University or City Hospitals in Italy, starting October 2006 and continuing until December 2010. The 100 patients randomised to the standard non PRO-CT guided antibiotic treatment plan will continue antibiotics for 10 days, whereas the 100 patients randomised to the PRO-CT-guided antibiotic treatment plan will continue for 10 days or stop antibiotics on day 3 depending on PRO-CT levels measured at admission, day 1 and day 2. Serum PRO-CT will be measured in a central laboratory. Patients will be examined at admission (visit 1), discharge and/or at 10 days (visit 4), 1 (visit 5), 3 (visit 6) and 6 months (visit 7). A telephone interview will be obtained at 2, 4 and 5 months. The primary outcome of the study will be the rate of exacerbations. Secondary outcomes will be hospital readmission, admission to ICU, change in FEV1, duration of hospitalization, and death. The sample size was estimated according to the primary outcome of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients who give written informed consent
* Age: adults >18 years old
* COPD diagnosis according to GOLD guidelines: FEV1/FVC <70% with FEV1<80% of predicted. If a COPD diagnosis is not evident from previous spirometric exams of the patient, a new spirometry will be obtained within 3 days of admission and a diagnosis of COPD will be made if all of the following conditions are true: 1) FEV1/FVC <70% with FEV1 <80% of predicted; 2) history of cigarette smoking; 3) exclusion of bronchial asthma diagnosis. At the end of the study (i.e. at 6 months) a new spirometric exam will be obtained from these patients to confirm the new diagnosis of COPD made at admission.
* Diagnosis of COPD exacerbation:

  * defined as acute-onset dyspnoea and/or cough associated with increased purulent sputum production (ANTHONISEN criteria)
  * requiring, according to guidelines (GOLD 2005), treatment with antibiotic
  * requiring hospitalization

Exclusion Criteria:

* Female subjects: pregnant, lactating mother or lack of efficient contraception in a subject with child-bearing potential (e.g. contraceptive methods other than oral contraceptives, IUD, tubal ligation)

  * Diagnosis of bronchial asthma
  * Coexisting medical conditions: unstable concomitant cardiovascular, renal, hepatic, gastrointestinal, neurological, endocrine, metabolic, muscle-skeletal, neoplastic, respiratory or other clinically significant disease (patients with stable and well controlled hypertension or diabetes may be included in the study)
  * Clinical significant laboratory abnormalities indicating unstable concomitant disease
  * Patients in whom survival for at least 1 year is unlikely
  * Inability to give informed consent

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of COPD according to GOLD guidelines
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2006-10; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo M Fabbri, MD, Principal Investigator — University of Modena and Reggio Emilia
Locations (1):
- University of Modena and Reggio Emilia, Modena, Italy

REFERENCES:
- [Derived] Verduri A, Luppi F, D'Amico R, Balduzzi S, Vicini R, Liverani A, Ruggieri V, Plebani M, Barbaro MP, Spanevello A, Canonica GW, Papi A, Fabbri LM, Beghe B; FARM58J2XH Study Group. Antibiotic treatment of severe exacerbations of chronic obstructive pulmonary disease with procalcitonin: a randomized noninferiority trial. PLoS One. 2015 Mar 11;10(3):e0118241. doi: 10.1371/journal.pone.0118241. eCollection 2015. PMID 25760346

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment process involved18 university/city hospital pulmonary departments. Patients selected were subjects hospitalized because of severe exacerbation of COPD (increased dyspnea, sputum volume, and sputum purulence according to Anthonisen criteria and/or respiratory failure) requiring antibiotic treatment.
Groups:
- PRO-CT Group: Experimental: COPD patients in the PRO-CT group will continue or discontinue antibiotic therapy depending on PRO-CT values.
  PRO-CT values: - continue antibiotics for 10 days if a single PRO-CT value is 0.25 mcg/L or greater, that will be judged suggestive of bacterial infection
  * continue antibiotics from day 3 to day 10 if one or more PRO-CT values are 0.1 to 0.25 mcg/L, indicative of possible bacterial infection, PLUS acute respiratory failure or clinical instability
  * stop antibiotics on day 3, if one or more PRO-CT values are between 0.1 to 0.25 mcg/L, indicative of possible bacterial infection, BUT the patient has not acute respiratory failure or clinical instability
  * stop antibiotics if all the PRO-CT values are < 0.1 mcg/L or if there is a consistent trend to normalization of PRO-CT with the last value < 0.1 mcg/L, that will be judged suggestive of absence of bacterial infection.
Period: Overall Study
Arm/Group | PRO-CT Group: Experimental | Standard Group: No Intervention
Started | 91 | 90
Completed | 88 | 90
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PRO-CT Group: Experimental | Standard Group: No Intervention | Total
Number analyzed (Participants) | 91 | 90 | 181
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Age, median (IQR)
  years | 73.5 [68.5 to 78] | 72.5 [65 to 78] | 73 [66.5 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 80 | 77 | 157
Region of Enrollment [Number; unit: participants]
  Italy | 91 | 90 | 181

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Rate of Severe Exacerbations in COPD, Comparing COPD Patients Previously Treated According to the PRO-CT Protocol Versus COPD Patients Previously Treated With Standard Antibiotic Therapy.
Description: We prospectively recruited COPD patients hospitalized for severe exacerbation of COPD and followed them after discharge. The primary end point of the study was the number of patients with at least 1 exacerbation at 6 months after the index exacerbation that was the reason for their hospital admission.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | PRO-CT Group: Experimental | Standard Group: No Intervention
Number analyzed (Participants) | 91 | 90
participants | 28 [-7.23 to 15.31] | 25 [-7.23 to 15.31]

2. Secondary Outcome: Cost/Effectiveness of the Use of PRO-CT-guided Decision Making Protocol on Duration of Antibiotic Therapy in COPD Exacerbations.
Time Frame: Discharge /10 days-6 months
Reporting Status: Not Posted

3. Secondary Outcome: To Evaluate if the PRO-CT-guided Decision Making to Shorten Antibiotic Therapy is Less Effective Than the Guideline Recommended Standard Antibiotic Treatment in Preventing Hospitalization.
Description: We evaluate the number of hospital re-admissions for severe COPD exacerbation in COPD patients of the study population, both in the PRO-CT group and in the standard group, in order to assess if shortening antibiotic therapy taking into account the values of PRO-CT is less effective compared to a standard antibiotic treatment.
Time Frame: Discharge/10 days-6 months
Reporting Status: Not Posted, anticipated posting 2014-11

4. Secondary Outcome: To Verify Survival in COPD Patients Comparing to Those Treated According to the PRO-CT Protocol Versus COPD Patients Treated With Standard Antibiotic Therapy.
Description: We evaluate the number of deaths from any cause among COPD patients in the study population, in order to compare survival among patients both in PRO-CT group and in the standard group.
Time Frame: Discharge/10 days-6 months
Reporting Status: Not Posted, anticipated posting 2014-11

5. Secondary Outcome: To Verify Changes in FEV1 Value in COPD Patients Comparing Those Treated According to the PRO-CT Protocol Versus COPD Patients Treated With Standard Antibiotic Therapy.
Description: COPD patients of the study population will undergo spirometry on visit 1, 4, 5, 7 in order to evaluate if there is change in FEV1 among COPD patients, both in the PRO-CT Group and in the standard Group.
Time Frame: Discharge/10 days-6 months
Reporting Status: Not Posted, anticipated posting 2014-11

6. Secondary Outcome: To Verify the Duration of Hospitalization for Severe Exacerbation in COPD Patients Treated According to the PRO-CT Protocol Versus COPD Patients Treated With Standard Antibiotic Therapy.
Description: We evaluate the duration in days in case of hospitalization for severe COPD exacerbation in COPD patients in the study population, both in the PRO-CT-guided antibiotic treatment group and in the standard antibiotic treatment group.
Time Frame: Discharge/10 days-6 months
Reporting Status: Not Posted, anticipated posting 2014-11

ADVERSE EVENTS:
Time Frame: 6 months after the index exacerbation
Arm/Group | PRO-CT Group: Experimental | Standard Group: No Intervention
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/90
Other Adverse Events (participants affected / at risk) | 0/91 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No